CLINICAL TRIAL: NCT02770326
Title: Safety of Fecal Microbiota Transplantation (FMT) for Recurrent or Refractory C. Difficile Infection in Patients With Solid Tumors
Brief Title: Safety of Stool Transplant for Patients With Difficult to Treat C. Difficile Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-337
Record Dates: First submitted 2016-05-11; First posted 2016-05-12 (Estimated); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2024-02

CONDITIONS: C. Difficile Infection; Cancer
Keywords: Safety of Stool Transplant; Fecal Microbiota Transplantation (FMT); 15-337
MeSH Terms: conditions — Neoplasms | interventions — Fecal Microbiota Transplantation

ARMS (1):
- Fecal Microbiota Transplantation (FMT) (Experimental): Patients with recurrent or refractory CDI who meet study eligibility criteria, will consent to undergo either colonoscopy or upper endoscopy with infusion of stool admixture. Safety will be assessed by monitoring infections that occurred within 2 weeks of the FMT procedures. Additionally, 24-hours, 1 week, 2 weeks, 4 weeks, and 6 months post-FMT, a stool sample will be collected. The time window for each time point listed is +/- 48 hours, with the exception of the first, 24 hour, time point. The time window for the 24 hour time point is +48 hours post FMT.
  Interventions: Biological: Fecal Microbiota Transplantation (FMT)

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation (FMT)

SUMMARY:
The purpose of this study is to test the safety of FMT in patients with C. difficile and cancer. In previous other studies, FMT has been shown to cure C. difficile when antibiotics have failed, but most of these studies have not included patients with cancer. The investigators want to prove that FMT is safe in this group of people so that doctors will feel more comfortable prescribing it for their patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Patients with solid organ malignancy who have received chemotherapy within the past six months.
* Clinical and microbiologic relapse of C. difficile associated diarrhea after at least one course of adequate antibiotic therapy or refractory disease that does not respond to treatment.

  * At least 10 days of vancomycin at least 125mg QID, or metronidazole 500mg TID
  * C. difficile associated diarrhea is defined as: ≥3 loose or watery stools per day for at least 2 consecutive days or ≥8 loose stools in 48 hours and Positive Clostridium difficile PCR
* Life expectancy of >3 months.

Exclusion Criteria:

* Expected prolonged compromised immunity

  * HIV infection with CD4 count <240
  * History of hematopoietic stem cell transplant (HSCT)
  * Hematologic malignancy
  * ANC <1000/mm3
* Contraindications to anesthesia for procedure

  * Serious cardiopulmonary comorbidities
  * Inability to tolerate anesthesia
  * HGB <8 g/dL
* Risk of bleeding during procedure

  * PLT <50,000 K/mcL
  * INR >1.5 INR
* Pregnancy

  o Pregnant patients will be excluded from this study.
* Gastrointestinal (GI) contraindications

  * Inflammatory bowel disease
  * Active fistula
  * Small bowel obstruction
  * Ileus
  * Gastroparesis
  * Nausea and vomiting
  * Gastrointestinal surgery within the previous 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-05-10 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin B. Mendelsohn, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Fecal Microbiota Transplantation (FMT): Patients with recurrent or refractory CDI who meet study eligibility criteria, will consent to undergo either colonoscopy or upper endoscopy with infusion of stool admixture. Safety will be assessed by monitoring infections that occurred within 2 weeks of the FMT procedures. Additionally, 24-hours, 1 week, 2 weeks, 4 weeks, and 6 months post-FMT, a stool sample will be collected. The time window for each time point listed is +/- 48 hours, with the exception of the first, 24 hour, time point. The time window for the 24 hour time point is +48 hours post FMT.
  Fecal Microbiota Transplantation (FMT)
Period: Overall Study
Arm/Group | Fecal Microbiota Transplantation (FMT)
Started | 10
Completed | 6
Not Completed | 4
Not completed — Death | 3
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Fecal Microbiota Transplantation (FMT)
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 67 [40 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Evaluated for Infection During Treatment Intervention
Description: Safety will be assessed by monitoring two types of infections that occur within 2 weeks of the FMT procedure.
Time Frame: 2 weeks after the FMT
Measure: Count of Participants; unit: Participants
Arm/Group | Fecal Microbiota Transplantation (FMT)
Number analyzed (Participants) | 10
Participants | 10

ADVERSE EVENTS:
Time Frame: 2 weeks after the FMT
Arm/Group | Fecal Microbiota Transplantation (FMT)
All-Cause Mortality (participants affected / at risk) | 7/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fecal Microbiota Transplantation (FMT) (N=10)
Anemia (Blood and lymphatic system disorders) | 10
Hypoalbuminemia (Metabolism and nutrition disorders) | 10
Hyperglycemic (Metabolism and nutrition disorders) | 8
Alkaline phosphatase increased (Investigations) | 7
Hypocalcemia (Metabolism and nutrition disorders) | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 6
Platelet count decreased (Investigations) | 6
White blood cell count (Investigations) | 6
Hypokalemia (Metabolism and nutrition disorders) | 5
Lymphocyte count decreased (Investigations) | 5
Neutrophil count decreased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 4
Activated partial thromboplastin time prolonged (Investigations) | 3
INR increased (Investigations) | 3
Blood bilirubin increased (Investigations) | 2
Creatinine increased (Investigations) | 2
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-25): https://cdn.clinicaltrials.gov/large-docs/26/NCT02770326/Prot_SAP_000.pdf